CLINICAL TRIAL: NCT02079051
Title: Impact of Medical Weight Loss on Physical Function in Severely Obese Older Adults
Brief Title: Impact of Weight Loss on Physical Function
Acronym: OPTIFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00025897
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Obesity Physical Performance Weight loss Optifast
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Weight Loss (Experimental): High intensity medical weight loss
  Interventions: Behavioral: High intensity medical weight loss
- Moderate Intensity Weight Loss (Active Comparator): Moderate intensity weight loss
  Interventions: Behavioral: Moderate intensity weight loss

INTERVENTIONS:
Behavioral: Moderate intensity weight loss — A calorie restricted diet based on estimates of total energy expenditure (TEE) obtained from the measured resting metabolic rate (RMR) during a wt stable period. TEE will be estimated by multiplying RMR by a factor of 1.1-1.3 to cover activity energy expenditure based on an assessment of physical activity levels at baseline using accelerometry. We will use the TEE to create an individualized dietary rx for each pt, subtracting up to 500 calories from the estimated TEE. To ensure micronutrient needs are being met, total calories will not be decreased below 1200 kcal per day, regardless of the estimated TEE. They will receive a standard exercise program that will be designed to promote exercise energy expenditure of approximately 1200 kcal/week. We will prescribe resistance training for 2 days per week with a loading intensity of 60% of 1 rep max and volume of 3 sets at 8 reps per exercise. Aerobic training will be prescribed for 3 days per week.
  Arms: Moderate Intensity Weight Loss
Behavioral: High intensity medical weight loss — Placed on complete meal replacement (MR) using the OPTIFAST medical wt loss protocol. Pts will consume a min of 86 g of protein daily in 5-6 servings of MR. Min caloric intake will be 960 kcal/day with adjustments in intake made based on BMI and activity levels, holding the percent of calories from protein constant at 35%. The MRs provide 100% of daily recommended needs for micronutrients and will be supplied weekly at clinic visits by the study. Pts will begin to incorporate food into their routine beginning at week 13 with guidance from a dietitian. From weeks 13-26, caloric prescriptions will be between 1100 to 1600 kcal/day, using a combo of MRs and food. Will receive an exercise program designed to promote exercise energy expenditure of approximately 1200 kcal/week. We will prescribe resistance training for 2 days per week with a loading intensity of 60% of 1 rep max and volume of 3 sets at 8 reps per exercise. Aerobic training will be prescribed for 3 days per wk.
  Arms: High Intensity Weight Loss

SUMMARY:
We are proposing a trial to directly compare a high intensity weight loss protocol to a moderate intensity weight loss protocol to determine which leads to greater improvements in physical function in severely obese older adults.

DETAILED DESCRIPTION:
We are proposing a trial to directly compare a high intensity weight loss protocol to a moderate intensity weight loss protocol to determine which leads to greater improvements in physical function in severely obese older adults. We are also interested in comparing the safety of the two approaches. If we can demonstrate effective weight reduction that happens with sufficient expediency and impact to improve physical functioning without increasing adverse events in severely obese older adults, a sizable percentage of the population would benefit and there would be significant reductions in disability resulting in cost savings for the healthcare system.

This application specifically addresses objective 3 as detailed in the announcement of this pilot funding mechanism (Objective 3. To develop and reliably test in clinical or pre-clinical studies novel interventions which target adiposity, peripheral or central nervous system, vascular, body composition and/or musculoskeletal related factors for preventing the age-related decline in physical function and preventing or reversing the progression to disability). This application describes a pilot randomized, controlled trial designed to address the following aims:

* Assess efficacy and safety of high intensity medical weight management in severely obese (= stage II BMI) older adults for functional outcomes (i.e., functional weight loss) compared to a moderate intensity weight loss intervention.
* Determine if a potential dose response relationship exists between weight loss volume (primarily as excess fat) and improvements in several measures of physical function.
* Identify changes in body composition (fat and lean including bone) that are associated with changes in physical function.
* Identify biomarkers (specific focus on markers of inflammation) that provide potential mechanistic links between weight reduction and changes in physical function in severely obese older adults.

Our primary hypothesis is that there is a greater improvement in physical function with a high intensity weight loss intervention compared to a moderate intensity intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old at the time of the initial screening visit
* BMI greater than or equal to 35 kg/m2

Exclusion Criteria:

* Cognitive impairment (Montreal Cognitive Assessment < 20)
* Depression (Centers for Epidemiologic Studies Depression Scale score >16
* Recent weight change (+/- 10 lbs. in the last 12 months)
* History of non-skin cancer in the last 2 years
* Cardiovascular disease event or unstable angina within the past six months, severe pulmonary disease, renal failure
* Major liver dysfunction within the last 2 years
* Recently quit smoking less than 12 months prior
* Use of estrogen or testosterone replacement therapy
* Current use of medications for psychosis or manic-depressive illness
* Use of weight-loss medications in previous 3 months
* Dependence on others for food procurement or preparation
* Poorly controlled diabetes (HgA1c greater than or equal to 9%) or blood pressure (greater than or equal to 159 mm Hg systolic or 99 mm Hg diastolic)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) | 6 months
  It is a measure of lower-extremity function consisting of walking speed, balance, and repeated chair stands. These 3 performance measures are scored from 0 to 4, with 4 indicating the highest level of performance and 0 the inability to complete the task. The summary score ranges from 0 (worst) to 12 (best). The SPPB is a well-studied composite measure and a strong predictor of disability, institutionalization, morbidity and mortality in initially non-disabled older persons. The reliability of the individual components, as well as the summary score, are good, with intra-class correlation coefficients above 0.88, and the measure is sensitive to change. Even small changes of 0.5-0.6 points have been shown to be clinically meaningful. Importantly, it has recently been advocated as an important primary outcome to be used in RCTs designed to develop evidenced-based interventions to prevent or postpone functional decline.

CONTACTS AND LOCATIONS:
Overall Officials: Jamy Ard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States